CLINICAL TRIAL: NCT05002920
Title: Correlation Between Body Mass Index and Progressive Bone Mineral Density in Cleft Patients After Secondary Alveolar Bone Grafting
Brief Title: Correlation Between Body Mass Index and Progressive Grafted Bone in Cleft Patients
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Pangyunchou, Assistant Professor, Chang Gung Memorial Hospital
Other Study IDs: 201702342A3C501
Record Dates: First submitted 2021-07-30; First posted 2021-08-12 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Cleft Lip and Palate; Bone Graft; Complications
Keywords: alveolar bone grafting; body mass index; bone mineral density; cone beam computed tomography
MeSH Terms: conditions — Cleft Lip | interventions — Alveolar Bone Grafting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cleft patients received alveolar bone grafting: alveolar bone grafting was performed when the cleft patients were aged around 9 years old. CBCT was used to analyze the bone mineral density of grafted tissue.
  Interventions: Procedure: alveolar bone grafting

INTERVENTIONS:
Procedure: alveolar bone grafting — the surgery of alveolar bone graft for alveolar defect in cleft patients

SUMMARY:
The cleft patients received alveolar bone graft(ABG) for alveolar defect. Body mass index (BMI) was measured for each patients when receiving ABG. Bone mineral density was measured by Cone-Beam CT at two time-points: post-ABG six months, and post-ABG two years. The study was to analyze the correlation between BMI and post-operative bone mineral density.

DETAILED DESCRIPTION:
Although childhood obesity is a growing issue, the association between BMI and the progressive bone mineral density (BMD) in grafted tissue after secondar alveolar grafting (ABG) remains little reviewed. This study compared the correlation between BMI and the progressive BMD after ABG procedure. Thirty-nine patients with unilateral or bilateral clefts were enrolled. ABG was performed at mixed-dentition age. Patient were classified into underweight, normal weight, and overweight or obese based on age- and sex-adjusted BMI. BMD was expressed in Hounsfield unit (HU) on cone-beam computed tomography (CBCT), which was obtained at 6 months (T1) and 2 years (T2) postoperatively. Calibrated BMD (HUgrafted tissue/HUpogonion¬, BMDc) was used for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* nonsyndromic unilateral or bilateral cleft lip and alveolus with or without palate patients
* received secondary ABG at Chang Gung Craniofacial Center
* received team managements based on our current treatment protocol for cleft lip and palate

Exclusion Criteria:

* syndromic cleft
* patients with failed grafted tissue

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: the patients with unilateral and bilateral cleft lip and palate received alveolar bone graft at their 9 year of age.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2021-01-25 (Actual); Primary Completion 2021-06-02 (Actual); Study Completion 2021-07-04 (Actual)

PRIMARY OUTCOMES:
bone mineral density | post-ABG six months
  measuring the bone density from cone beam CT
bone mineral density | post-ABG two years
  measuring the bone density from cone beam CT

CONTACTS AND LOCATIONS:
Overall Officials: Pangyun Chou, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
no plan shared.